CLINICAL TRIAL: NCT03668912
Title: Feasibility of a Guided Participation Discharge Program for Very Preterm Infants
Brief Title: Guided Participation Discharge Program for Very Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Lee Suk Yin, Principal Investigator, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2018-09-11; First posted 2018-09-13 (Actual); Last update posted 2018-09-14 (Actual); Status verified 2018-09

CONDITIONS: Very Premature Baby

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guided participation group (Experimental)
  Interventions: Behavioral: Guided participation discharge programme
- Usual care group (No Intervention)

INTERVENTIONS:
Behavioral: Guided participation discharge programme — A nurse-led GP discharge intervention (3 structured 30- to 60-minute GP sessions and 1 follow-up phone call)
  Arms: Guided participation group

SUMMARY:
This study aimed at investigating the feasibility of a new guided participation (GP) discharge program for parents of very preterm infants. A randomized controlled trial was conducted in a neonatal intensive care unit. The intervention included three structured GP sessions and one follow-up phone call. The control group received usual care. Outcomes measured included parents' efficacy and satisfaction with parenting, and perceived stress. Data collection was conducted at baseline, on day of discharge, after the follow-up phone call, and 1 month after discharge. The outcomes were analyzed on the basis of intention-to-treat principles.

ELIGIBILITY:
For Infants:

Inclusion Criteria:

- A gestational age of ≤32 weeks at birth

Exclusion Criteria:

* Have congenital malformation(s)
* Need to undergo a major surgery

For Parents:

Inclusion Criteria:

- Must be the infant's primary caregiver

Inclusion Criteria:

- Diagnosed with a mental illness

Max Age: 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Parents' change in score of Parenting Sense of Competence Scale from baseline to up to 8 weeks | Baseline, and at 3-, 4-, and 8-weeks after baseline
  The Chinese version of the Parenting Sense of Competence Scale is a self-reported instrument which includes 17 items in two subscales (efficacy and satisfaction). Each item is rated on a 6- point Likert scale ('Strongly disagree' = 1; 'Strongly agree' = 6). Nine items (items 2, 3, 4, 5, 8, 9, 12, 14 and 16) were reverse-coded. The total scores ranged from 17 to 102. A higher score indicates a higher sense of competence and satisfaction with parenting by parents.

SECONDARY OUTCOMES:
Parents' change in score of Perceived Stress Scale from baseline to up to 8 weeks | Baseline, and at 3-, 4-, and 8-weeks after baseline
  The Chinese version of the Perceived Stress Scale consists of 10 items. Each item is rated on a 5-point Likert scale ('never' = 0; 'very often' = 4). The total score is yielded by summing the scores of all items. The total score ranges from 0 to 40. The higher the score, the higher is the parents' perceived stress in parenting.

CONTACTS AND LOCATIONS:
Overall Officials: lsy307@ha.org.hk Lee, Principal Investigator — Department of Pediatrics, Prince of Wales Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee SY, Chau JPC, Choi KC, Lo SHS. Feasibility of a guided participation discharge program for very preterm infants in a neonatal intensive care unit: a randomized controlled trial. BMC Pediatr. 2019 Nov 4;19(1):402. doi: 10.1186/s12887-019-1794-y. PMID 31684903